CLINICAL TRIAL: NCT05689190
Title: Non-invasive Flow Measurements in Patients With Lower Extremity Arterial Disease (LEAD)
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000115
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lower Extremity Arterial Disease
Keywords: blood flow measurements

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Duplex ultrasound, angiogram, PTA intervention

SUMMARY:
This concerns a study with patients who will undergo endovascular treatment. Blood flow will be measured by 2D Duplex Ultrasound. Contrast data will be collected that will be processed offline.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the vascular surgery outpatient clinic (LUMC) with PAD
* Age ≥18 years
* Superficial femoral artery (SFA) stenosis (>70% occluded)
* Elective for a percutaneous transluminal angioplasty procedure
* Written informed consent

Exclusion Criteria:

* Contraindications to angiography, such as severe renal insufficiency (eGFR< 20)
* Non-correctable bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients that are referred to the Vascular Surgery outpatient clinic (department of Vascular Surgery) with PAD and an indication for a percutaneous transluminal angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
blood flow | performed during a regular PTA intervention
  Repeatability and correlation of angiographic hemodynamic measurements compared with the golden standard 2D duplex ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Carla SP van Rijswijk, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No